CLINICAL TRIAL: NCT06875102
Title: Fatigue in Sjögren's Syndrome: a Randomized Controlled Trial of Combined Non-pharmacological Therapeutic Strategies
Brief Title: Fatigue in Sjögren's Syndrome: 3 Therapeutic Strategies
Acronym: FESSONA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24CH125; ANSM (Other: 2024-A02116-41)
Record Dates: First submitted 2025-02-04; First posted 2025-03-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Sjogren Syndrome
Keywords: Sjögren's Syndrome; fatigue; acupuncture; adapted physical activity (APA); transcutaneous vagal nerve stimulation (tVNS)
MeSH Terms: conditions — Sjogren's Syndrome; Fatigue | interventions — Acupuncture Therapy; Glutamyl Aminopeptidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- APA + sham ACU + tVNS (Experimental)
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation (tVNS); Other: APA (adapted physical activity ); Device: Acupuncture (sham_ACU)
- APA + ACU + simulated tVNS (Experimental)
  Interventions: Device: Acupuncture (ACU); Other: APA (adapted physical activity ); Device: Simulated Transcutaneous Vagus Nerve Stimulation (sim_tVNS)
- APA + Simulated tVNS + sham ACU (Sham Comparator)
  Interventions: Other: APA (adapted physical activity ); Device: Acupuncture (sham_ACU); Device: Simulated Transcutaneous Vagus Nerve Stimulation (sim_tVNS)

INTERVENTIONS:
Device: Acupuncture (ACU) — acupoints will be Baihui (GV20); Zhongwan (CV12), Guanyuan (CV4), bilateral Zusanli (ST36) bilateral Taichong (LV3). The needles will remain for 30 min. Subjects will receive acupuncture twice a week during the 12-week intervention.
  Arms: APA + ACU + simulated tVNS
Device: Transcutaneous Vagus Nerve Stimulation (tVNS) — Transcutaneous Vagus Nerve Stimulation (tVNS) will be performed using an ECO TENS 2 device with an ear clip put in the conque aurea of the left ear, which is innervated by the auricular branch of the vagus nerve. In the groups receiving simulated tVNS, stimulation will be delivered to the ear lobe, which is devoid of vagal innervation.
  Stimulation will be delivered at a frequency of 20 Hz and a pulse width of 200 ms, while the stimulation amplitude will be individually titrated to 1 mA below the level that will lead to a mild unpleasant feeling, according to the parameters defined by Stavrakis et al (2017, 2020).
  Arms: APA + sham ACU + tVNS
Other: APA (adapted physical activity ) — The APA (adapted physical activity ) program : 2 sessions of 90 min (with 60 min of aerobic exercise and 30 min of resistance exercises per session) per week, for 12 consecutive weeks
Device: Acupuncture (sham_ACU) — Needles well be used in the non-acupoint area 2 centimeters away from the real acupoints. The needles will remain for 30 min. Subjects will receive sham acupuncture twice a week during the 12-week intervention.
  Arms: APA + Simulated tVNS + sham ACU; APA + sham ACU + tVNS
Device: Simulated Transcutaneous Vagus Nerve Stimulation (sim_tVNS) — Simulated Transcutaneous Vagus Nerve Stimulation (sim_tVNS) will be performed using an ECO TENS 2 device with an ear clip put in the conque aurea of the left ear, which is innervated by the auricular branch of the vagus nerve. NSVt devices will be used in "simulated" mode.
  Arms: APA + ACU + simulated tVNS; APA + Simulated tVNS + sham ACU

SUMMARY:
Unexplained fatigue is a frequent (60-70%) chronic complaint in Sjögren's syndrome (SjS) with a clear unmet therapeutic need, despite the recommendation of adapted physical activity (APA) programs, which are effective and feasible, but only to some extent. Hence, other therapeutic approaches, such as Acupuncture (ACU) or transcutaneous vagal nerve stimulation (tVNS), have been evaluated during the past years, with varying degrees of success in alleviating fatigue.

FESSONA has been designed as a randomized controlled monocentric trial, aiming at comparing the effects of 3 different programs on fatigue in SjS: APA alone, APA+ACU and APA+tVNS. Relevant controls will be included as well (sham ACU and simulated tVNS).

Multiple fatigue and SjS-related features will be measured before (at inclusion) and after (week 12) the intervention, as well as at week 24 and 48, to evaluate the short- and long-term impact of each program. Tolerance and feasibility will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security scheme.
* Age > 18 years.
* Patient informed and having signed the information form and consent to participate in the study.
* Patient with Sjögren's syndrome according to ACR/EULAR 2016 or AECG 2002 criteria, usually followed up every year or more frequently
* Fatigue present for ≥ 6 months, without obvious explanation and/or specific treatment to conduct (e.g., disease's flare, chronic infection), with a current FACIT-F score < 34

Exclusion Criteria:

* Pre-existing atrial fibrillation or severe cardiac conduction disorders,
* Recent stroke or myocardial infarction (<6 months),
* Left ventricular ejection fraction <40% or severe heart failure (New York Heart Association functional class III or IV)
* Recurrent episodes of vasovagal syncope, or history of vagotomy
* People with dermatological problems in the area where the stimulation electrodes are to be placed
* Current episode of venous or arterial thrombosis
* Pregnancy or breastfeeding
* Patient under protective measures (legal protection, curatorship, guardianship)
* Inability or refusal to understand and/or sign informed consent to participate in the study, or to perform follow-up examinations required under the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue score assessed | Between inclusion (week 0) and visit V1 at 12 weeks (± 1 week from the end of the 12-week program)
  Change in fatigue score assessed using the FACIT-F questionnaire (Functional Assessment of Chronic Illness Therapy - Fatigue; ranging from 0 to 52, 0 meaning extreme fatigue and 52 the total absence of fatigue)

SECONDARY OUTCOMES:
FACIT-F score in the different groups | between inclusion (Week 0) and week 48
  FACIT-F score at 48 weeks, in the different groups
Root Mean Square of the Successive Differences in heart rate or RMSSD (in milliseconds) | at 12, 24 and 48 weeks,
  Root Mean Square of the Successive Differences in heart rate or RMSSD (in milliseconds), measured from a nocturnal ECG recording by Holter ECG, in the different groups
Proportion (in %) of the 24 APA sessions carried out (at least 80% of the exercises proposed) in the different groups | week 48
ClinESSDAI score | at 12, 24 and 48 weeks,
  ClinESSDAI score (clinical part of the EULAR Sjögren's Syndrome Disease Activity Index; assessed on 11 "domains" corresponding to the main clinical manifestations of the disease; ranging from 0 to 135, a score of 0 meaning the existence of a disease and a score of 135 a disease whose activity would be maximal) in the different groups
ESSPRI questionnaire (EULAR Sjögren's Syndrome Patient Reported Index) | at 12, 24 and 48 weeks
  ESSPRI questionnaire (EULAR Sjögren's Syndrome Patient Reported Index); calculated as the mean of 3 self-measurement scales assessing fatigue, dryness and pain, each ranging from 0 to 10; 0 meaning the total absence of the symptom considered and 10 a symptom whose intensity would be at the maximum imaginable) in the different groups
HADS questionnaire (Hospital Anxiety and Depression Scale) | at 12, 24 and 48 weeks
  HADS questionnaire (Hospital Anxiety and Depression Scale) composed of an anxiety score and a depression score both ranging from 0 to 21, 0 meaning the absence of symptoms of this type, and 21 the presence of an anxiety and/or major depressive state) in the different groups
Self-measurement questionnaire SF-36 (Short Form Health Survey 36) | between inclusion (Week 0) and week 48
  Self-measurement questionnaire SF-36 (Short Form Health Survey 36); comprising 36 questions assessing 8 dimensions, namely physical functioning, role limitation due to physical problems, role limitation resulting from emotional problems, vitality (energy/fatigue), emotional well-being, social functioning, bodily pain, and perception of general and mental health; each dimension is represented by a score ranging from 0 to 100, with a low score signifying poor health perception in the dimension considered, and a high score signifying the opposite)
EQ-5D-5L self-measurement questionnaire assessing 5 dimensions of health | at 12, 24, and 48 weeks,
  EQ-5D-5L self-measurement questionnaire assessing 5 dimensions of health (mobility, autonomy, daily activities, pain/discomfort and anxiety/depression) with 1 question per domain, with the possibility of choosing 5 degrees of severity each time (1 corresponding to no difficulty for the domain and 5 corresponding to the maximum degree of difficulty in the domain), the total of the 5 notes of the 5 domains giving a score ranging from 5 to 25, and this questionnaire is associated with a visual analogue scale (VAS) allowing the patient to rate his state of health of the day from 0 (the worst state of health imaginable) to 100 (the best state of health imaginable), in the different groups
Schirmer test | at 12, 24 and 48 weeks
  the area of the graduated blotter that became wet after 5 min of placement on the lower eyelid of each eye, expressed in millimeters and as the average of the two eyes) at 12, 24 and 48 weeks, in the different groups
VO2max | at 12, 24 and 48 weeks
  VO2max (in ml/min/kg; after metabolic test) in the different groups
Handgrip test | at 12, 24 and 48 weeks
  Handgrip test (in kg; via a grip test on the dominant upper limb) in the different groups
Number of daily steps | at 12, 24 and 48 weeks
  Number of daily steps measured via a connected watch on average over the week preceding the assessments at 12, 24 and 48 weeks, in the different groups

CONTACTS AND LOCATIONS:
Overall Officials: Martin KILLIAN, MD, Principal Investigator
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou X, Chen J, Colas C, Hupin D, Killian M. FatiguE in Sjogren's Syndrome: a randomised controlled trial of cOmbined Non-phArmacological therapeutic strategies (FESSONA). BMJ Open Sport Exerc Med. 2025 Jun 16;11(2):e002677. doi: 10.1136/bmjsem-2025-002677. eCollection 2025. PMID 40546749